CLINICAL TRIAL: NCT06118580
Title: Aggression and Social-Emotional Information Processing: Neural Correlates During Alcohol Intoxication.
Brief Title: Neural Correlates During Alcohol Intoxication
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Emil Coccaro, Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2020H0369
Record Dates: First submitted 2023-11-01; First posted 2023-11-07 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Alcohol Use Disorder; Intermittent Explosive Disorder
Keywords: AUD; IED; Social Cognition
MeSH Terms: conditions — Alcoholism; Disruptive, Impulse Control, and Conduct Disorders | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Placebo drink (without alcohol)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oral alcohol drink (Experimental)
  Interventions: Drug: Alcohol (Ethanol)
- Placebo (non-alcohol drink) (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Alcohol (Ethanol) — 95% Ethanol diluted in Grape-flavored drink
  Arms: Oral alcohol drink
Drug: Placebo — Grape-flavored drink
  Arms: Placebo (non-alcohol drink)

SUMMARY:
Alcohol intoxication is responsible for a large proportion of violent crime/assault and personal injury in our society. While a number of variables have been associated with alcohol-related aggression, high trait aggression and impaired executive function have been identified as key factors. Both Alcohol Use Disorder (AUD) and Impulsive Aggression behavior (AGG) are related to impaired social-emotional information processing (SEIP) whereby social threat cues, especially ones that are ambiguous in nature, lead to hostile attribution and negative emotional response to the "other" and, then, aggression against the "other". Thus, understanding the underlying neuroscience of SEIP under the influence of alcohol will be critical to identifying targets for intervention to reduce alcohol-related aggressive behavior. In addition to potential pharmacologic and cognitive-behavioral based interventions, such interventions may also involve the rehabilitation of aberrant neuronal circuits underlying social cognitive function through neuroplasticity-based remediation exercises. This study is designed to see how brain activation of cortico-limbic circuits involving social-emotional information processing, analyzed by fMRI Imaging, are impacted by alcohol administration in those with and without aggressive disorders and with and without alcohol use disorder.

DETAILED DESCRIPTION:
A critical issue related to aggression and to alcohol-related aggression is the role of social-emotional information processing (SEIP) including hostile attribution bias (HAB). SEIP can explain the development and maintenance of impulsive aggressive behaviors. SEIP involves a multi-stage set of processes involving (1) encoding of social information, (2) attribution of the intent of the behavior of the other participant, and (3) emotional response. Ultimately, deficits in SEIP lead to aggressive behavior because the misperception of emotional stimuli in social encounters leads to hostile attribution, anger, and then, an inappropriate aggressive response. Experimental studies consistently demonstrate that acute intake of alcohol facilitates aggressive behavior. These studies have typically measured aggression with the Taylor Aggression Paradigm (TAP) in which aggression occurs in the context of electric shocks to a fictitious opponent in response to electric shocks that this opponent gives to the subject during a reaction-time task. Generally, individuals who receive alcohol respond more aggressively (i.e., set higher shocks) than those who receive a non-alcoholic placebo beverage. Importantly, these studies report that provocation is a necessary component for aggressive behavior to occur during alcohol intoxication. Simply put, alcohol-induced aggression is elicited when participants are provoked. Other relevant factors in alcohol-related aggression include impairments in executive cognitive function (ECF) and disruption of cognitive processes critical for self-regulation (e.g., attention, inhibition, information processing, and decision making), all of which are important in social-emotional information processing (SEIP). In fMRI studies, during alcohol infusion, decreased responses were observed in cortical areas [anterior cingulate cortex (ACC) and in the dorsomedial PFC (dmPFC)], and increased responses in subcortical areas [AMYG and ventral striatum (VS)]. In addition, increases in responses in AMYG and in VS were both correlated with aggressive responding to provocation during the TAP test. Emerging data indicate that acute alcohol intoxication alters cortico-limbic circuits in healthy, non-alcoholic, individuals and that history of alcoholism or aggression also alters these circuits.

ELIGIBILITY:
Inclusion Criteria:

1. Inclusion Criteria for All Participants: All candidates for this study must meet the following criteria:

   1. 21 to 55 years of age (and be righted handed) and not a current (past 3 months) alcohol abstainer.
   2. Consumes > 10 drinks/week or reports binge drinking at least once a month, and is not in, or currently seeking, treatment for AUD.
   3. PCL-SV psychopathy score < 18
   4. Able/willing to abstain from alcohol for 24 hours before MRI scanning.
   5. Physically healthy (confirmed by comprehensive medical history and physical exam) and does not have metal implants, plates, or screws in body or head (MRI safety issue).
   6. If a smoker, consumes no more than 15 cigarettes per day.
   7. Able to give informed consent.
2. Inclusion Criteria for AGG (Only) Participants: In addition to the above, all AGG candidates must meet the following criteria:

   1. Life History of Aggression (LHA) score > 12
   2. In addition AGG participants must report:

      1. Current history of at least two (2) angry outbursts a week (on average) for the past three months and/or three significant angry aggressive outbursts in which other people are assaulted and/or property is damaged in the past year.
      2. Angry outbursts are out of proportion to provocation and not associated with a tangible goal (not premeditated).
      3. Angry outbursts are associated with distress and/or impairment;
      4. Angry outbursts do not occur exclusively during another disorder or condition.
   3. No lifetime history of AUD (from DSM-5 criteria).
3. Inclusion Criteria for AUD (Only) Participants: In addition to the above, all AUD candidates must meet the following criteria:

   1. Meets DSM-5 criteria for alcohol use disorder (AUD) without significant history of alcohol withdrawal, seizures, or delirium tremens.
   2. Consumes > 10 drinks/week or reports binge drinking at least once a month, and is not in, or currently seeking, treatment for AUD.
4. Inclusion Criteria for AUD+ / AGG+ Participants: These participants meet criteria for both AUD and AGG as described above.
5. Inclusion Criteria for Non-AGG/Non-AUD (Healthy Control) Participants: All Non-AGG/Non-AUD candidates must meet the following criteria:

   1. Does not meet DSM-5 criteria for current or past alcohol use disorder (AUD).
   2. LHA score is less than 12.
   3. Does not meet DSM-5 Criteria for a current, or past, major psychiatric disorder.

   b. Study Exclusion Criteria:

1) < 21 years of age or > 55 years of age. 2) Meets criteria for other (Non-AUD) current DSM-5 Substance Use Disorder (excluding tobacco use disorder provided the participant consumes no more than 15 cigarettes per day).

3) Life history of bipolar disorder, schizophrenia, organic mental syndrome or intellectual deficiency (i.e., IQ < 70 by WRAT).

4) Drug screen positive for amphetamines, barbituates, benzodiazepines, cocaine, phencyclidine, or opiates.

5) Positive urine pregnancy test 6) Clinically significant medical condition (current and active medical condition requiring daily prescribed medication).

7) PCL-SV psychopathy score > 18 (see above). 8) Score > 8 on the Clinical Institute Withdrawal Assessment-Revised (CIWA-Ar).

9) Treatment with antipsychotic medications within two weeks of study entry. 10) Current suicidal ideation. 11) Metal in body, history of > 5 min loss of consciousness, left-handedness or body weight > 300lbs (fMRI exclusions).

12) Unable/unwilling to abstain from alcohol for 24 hours and recreational drugs for 48 hours prior to session arrival.

13) Unable to comply with study procedures. 14) Unable to sign informed consent document. 15) Taking of anticoagulants. 16) Drinks less than 2 drinks per week 17) Has not had a binge drinking episode (5+ for men, 4+ for women) in the past 3 months.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 144 (Estimated)
Dates: Start 2023-06-08 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Cortico-limbic Response to Anger Faces | 60-120 minutes after Ethanol (or Placebo) drink
  Orbito-frontal and Amygdala responses to Anger Faces
Brain Connectivity | 60-120 minutes after Ethanol (or Placebo) drink
  Resting State

CONTACTS AND LOCATIONS:
Overall Officials: Emil Coccaro, M.D., Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No